CLINICAL TRIAL: NCT04077684
Title: Efficacy and Safety of Low-dose Interleukin-2 in Patients With Systemic Lupus Erythematosus: a Multicenter, Randomised, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Low-dose IL-2 in Patients With SLE: a Multicenter, Randomised, Placebo-controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Dept. Rheumatology and Immunology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018PHB041-01
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): placebo s.c. injection every other day for the first 12 weeks and then once a week for the second 12 weeks
  Interventions: Drug: Interleukin-2
- IL-2 at 0.2MIU (Active Comparator): 0.2 MIU doses of IL-2 s.c. injection every other day for the first 12 weeks and then once a week for the second 12 weeks
  Interventions: Drug: Interleukin-2
- IL-2 at 0.5MIU (Active Comparator): 0.5 MIU doses of IL-2 s.c. injection every other day for the first 12 weeks and then once a week for the second 12 weeks
  Interventions: Drug: Interleukin-2
- IL-2 at 1.0MIU (Active Comparator): 1.0 MIU doses of IL-2 s.c. injection every other day for the first 12 weeks and then once a week for the second 12 weeks
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — IL2 (0.2 MIU, 0.5 MIU or 1 MIU) : placebo = 1:1:1:1
  Other Names: Human recombinant IL-2

SUMMARY:
The management of active systemic lupus erythematosus (SLE) is challenging due to the heterogeneous nature of the disease and lack of specific treatment. Current treatment regimens mainly rely on corticosteroids and immunosuppressive agents which are associated with substantial adverse effects including various infections. Therefore, there is an unmet need for new therapies with better efficacy and less adverse effects.

Defective IL-2 production contributes to the unbalanced immune system in SLE. Previous short term open-labelled trials showed that low-dose IL-2 was efficient and tolerated in active SLE. It was suggested that low-dose IL-2 treatment promoted regulatory T cells (Treg) and inhibited T helper 17 cells (Th17) and follicular helper T cells (Tfh). The immunological rebalancing was associated with the induction of remission in SLE patients.

To establish that which low doses of IL-2 would be more efficacious and safe in active SLE, we carried out a multi-center, randomized, double-blind, placebo-controlled trial of three doses of IL2 (0.2 MIU, 0.5 MIU or 1 MIU) versus placebo.

DETAILED DESCRIPTION:
Active SLE patients at 18 to 75 years of age were enrolled. Patients were randomly assigned (in a 1:1:1:1 ratio) to one of the four arms (placebo or IL-2 at 0.2 MIU, 0.5 MIU or 1 MIU) in the study. IL-2 (0.2 MIU, 0.5 MIU or 1 MIU) or placebo was administered subcutaneously every other day for the first 12 weeks , and then was adjusted to once a week for the second 12 weeks. Follow-up visits occurred on weeks 4, 8,12,16,20 and 24. The end points were safety and clinical and immunologic response.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 1997 revised classification criteria of the American College of Rheumatology
2. SLE disease activity index(SLEDAI) ≥ 8
3. age:18 to 75 years, weight 45-80Kg
4. Patients had an inadequate response to standard treatment for ≥ 3 months. The background treatment included corticosteroids (≤1.0 mg/kg), hydroxychloroquine, cyclophosphamide , mycophenolate mofetil or other immunosuppressants.
5. Negative urine pregnancy test
6. Written informed consent form

Exclusion Criteria:

1. allergic to IL-2, corticosteroids, hydroxychloroquine, cyclophosphamide or mycophenolate mofetil
2. active severe neuropsychiatric manifestations of SLE;
3. hepatic insufficiency (alanine aminotransferase or aspartate aminotransferase ≥ 2 times of the upper limit of the normal range);
4. pregnancy or lactation in females.
5. Cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or Basocellular carcinoma);
6. Serious infection such as bacteremia, sepsis;history of chronic infection;
7. active infection (hepatitis B or C virus, Epstein-Barr virus, human immunodeficiency virus or Mycobacterium tuberculosis);
8. history vision and visual field disorders, cataract；
9. severe comorbidities including heart failure (≥ grade III NYHA)
10. active peptic ulcers；
11. complicated with other autoimmune diseases;
12. History of administration of rituximab or other biologics within 6 months;
13. therapy with other immunosuppressors;
14. participate in other clinical trial within 4 weeks;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
the response measured by the SLE Responder Index-4 (SRI-4) | week 12
  SRI response was defined as (1) a ≥ 4-point reduction in SELENA-SLEDAI score, (2) no new BILAG A score or ≤ 1 new BILAG B score, and (3) no deterioration from baseline in the physician's global assessment by ≥ 0.3 points.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheumatology and Immunology
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No